CLINICAL TRIAL: NCT07115849
Title: Effect of Different Sex Hormone Profiles for the Response to Physical Training
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Principal Investigator, Mette Hansen, Associate Professor, University of Aarhus
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 1-10-72-170-24
Record Dates: First submitted 2025-08-04; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Eumenorrhea; Intrauterine Devices, Medicated; Hormonal Contraception
Keywords: IUD; POPs; Progestin; sex hormone profile; physical training
MeSH Terms: interventions — Physical Conditioning, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Non-hormonal contraception users (Active Comparator): Non-hormonal contraception users
  Interventions: Behavioral: Physical training
- IUD users (Experimental): IUD users
  Interventions: Behavioral: Physical training
- Progestin only pill users (Experimental): Progestin only pill users
  Interventions: Behavioral: Physical training

INTERVENTIONS:
Behavioral: Physical training — Aerobic and resistance training three times per week. Two supervised training sessions.

SUMMARY:
The aim of the project is to elucidate the impact of diverse sex hormone profiles on the adaptability of muscle mass to physical training. Additionally, the project aims to investigate secondary effects on adipose tissue, tendons, and other physiological parameters associated with physical function.

DETAILED DESCRIPTION:
The human study is designed as a prospective study where 3 groups with different sex hormonal profiles are followed in parallel in 4 months and tested before, during (2 months) and after 4 months of physical training intervention. The three groups include a control group with regular menstrual bleeding and two groups who have an altered sex hormonal profile due to use of either IUD (containing the progestin levonorgestrel) or mini pills (containing the progestin desogestrel). Before and after the training period the following will be measured/collected: Body composition, Dietary intake, Physical Activity Level, Blood, Urine, Muscle Tissue, Adipose Tissue, Aerobic capacity in bike test, Strength and muscle function tests, and questionnaires about diet and physical activity.

ELIGIBILITY:
Inclusion Criteria:

* BMI 19-25

Exclusion Criteria:

* Training more than 2 times per week
* Smoking
* Pregnancy
* Taking any medications known to affect the outcome parameters

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-05 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Muscle mass | 4 months
  Muscle mass measured by DXA
Fat free mass | 4 months
  Fat free mass measured by DXA

SECONDARY OUTCOMES:
Muscle fiber | 4
  Muscle fiber type and area
Protein synthesis and degradation | 4 months
  Muscle protein synthesis and degradation
Adipose tissue sex hormone receptors | 4 months
  Adipose tissue sex hormone receptors
Resting metabolic rate | 4 months
  Resting metabolic rate measured via indirect calorimetry
Maximal oxygen uptake | 4 months
  Maximal oxygen uptake
Muscle strength | 4 months
  Muscle strength (arm and finger strength)
Appetite regulatory markers | 4 months
  Leptin, Ghrelin, CCK, GLP-1
Lipid profile | 4 months
  Lipid profile